CLINICAL TRIAL: NCT06817837
Title: Feasibility Study: The Contribution of Hypnosis in the Management of Adults With Brain Injuries
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Principal Investigator, Helena Cassol, Principal Investigator, Centre Hospitalier Universitaire de Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-446
Record Dates: First submitted 2025-01-28; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Stroke; Traumatic Brain Injury
Keywords: hypnosis; stroke; traumatic brain injury; pain; sleep disorders; anxiety; behaviorals disorders
MeSH Terms: conditions — Stroke; Brain Injuries, Traumatic; Pain; Sleep Wake Disorders; Anxiety Disorders | interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: An experimental group and a control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hypnosis (Experimental): The patients in the experimental group will receive 8 hypnosis sessions, scheduled one session every two weeks. These will replace one neuropsychology session for the patient (patients will still be followed in neuropsychological rehabilitation). The procedure will therefore last 4 months. These hypnosis sessions aim to address anxiety, sleep disorders, pain, and/or behavioral disorders.
  Interventions: Behavioral: hypnosis
- control (No Intervention): The patients in the control group will continue their usual multidisciplinary care without any changes.

INTERVENTIONS:
Behavioral: hypnosis — Eight hypnosis sessions will be offered to address various issues: sleep disorders, behavioral issues, anxiety, and pain.
  Arms: hypnosis

SUMMARY:
This controlled and randomized study aims to explore the feasibility and benefits of hypnosis in the management of patients who have suffered a traumatic brain injury or a stroke, by assessing its impact on behavioral disorders related to the dysexecutive syndrome, as well as associated symptoms (anxiety, sleep disorders, and pain).

For this study, a convenience sample of 40 adult patients with acquired brain injuries will be recruited and randomly assigned to two groups: one group will receive hypnosis sessions integrated into their usual care, and the control group will receive only conventional treatment. These patients are currently being followed in neurological rehabilitation with complaints (anxiety, sleep, pain, and/or behavioral disorders). These complaints will be initially assessed using visual analog scales (VAS) for these four points. Patients with scores higher than 4 on at least two of the scales will be admitted to the study. They will be randomly assigned to either the control or experimental group.

Sociodemographic data (age, sex, education) and certain medical data related to the brain injury will be collected, such as: the initial Glasgow Coma Scale score, medication treatment, lesion type, and the timing of the injury.

Several questionnaires and scales will be completed at patient inclusion and at the end of the protocol. The severity of behavioral disorders will be assessed using the DysEXecutive (DEX) questionnaire from the Behavioral Assessment of the Dysexecutive Syndrome (BADS). For anxiety, pain, and/or sleep disorders, the following questionnaires will be used: the State-Trait Anxiety Inventory (STAI), the Beck Depression Inventory, the Pittsburgh Sleep Quality Index (PSQI), and the Medical Outcome Study Short Form (SF-36) for quality of life.

For the hypnosis protocol (experimental group), 8 individual sessions will be offered to the patient, each lasting about one hour and spread over a period of 4 months (one hypnosis session every two weeks). The sessions will proceed as follows:

* In the first session, a history will be taken to gather the patient's request or issue for which they were referred for hypnosis, and specific goals will be established. An explanation of hypnosis will also be provided.
* The second session will offer a "safe haven" hypnosis, where the patient revisits a happy moment to find calm and a secure place.
* In the third session, a "red balloon" hypnosis will be offered, using a metaphor where the patient releases bothersome emotions.
* The fourth session will focus on sleep (hypnotic metaphor for sleep induction).
* The fifth session will use "object-tool" hypnosis, where the patient works on a specific issue represented metaphorically by an object and enhances it with tools that can modify it.
* The sixth session will introduce self-hypnosis training for the patient.
* The final two sessions will be personalized and address the patient's current needs.

At the end of each session, patients will be asked to complete a visual analog scale (VAS) to measure their level of absorption in the hypnosis.

Note that, except for the first two sessions, the order of the sessions may be slightly adjusted based on the patient's needs or requests. Patients in the control group will also complete the same questionnaires at inclusion and after 4 months.

During the 4-month period, all patients, from both the hypnosis and control groups, will continue to receive multidisciplinary rehabilitation care. Furthermore, the hypnosis sessions will replace one neuropsychology session each time so that both groups (control vs. hypnosis) receive the same number of sessions over the period. Finally, data will be analyzed for patients who have completed at least 80% of the prescribed hypnosis sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older;
* Acquired brain injury of the type stroke (AVC) or traumatic brain injury (TBI), regardless of the severity;
* Presence of complaints of anxiety, sleep disorders, disabling pain, and/or behavioral disturbances;
* Stability of medication treatment during the month prior to inclusion.

Exclusion Criteria:

* Patients already receiving hypnosis treatment or practicing hypnosis. Patients with prior experience with hypnosis before the injury may be included;
* Patients presenting or who have presented with aphasia;
* Patients still experiencing post-traumatic confusion;
* Patients with a history of psychiatric disorders;
* History of alcoholism or drug addiction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-05 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Short Form Health Survey (SF 36) | At the inclusion of the patient and up to 8 weeks
  This is a self-reported questionnaire designed to assess health-related quality of life. It includes 36 items distributed across 8 dimensions: physical function, physical role limitations, bodily pain, general health, vitality, social function, emotional role limitations, and mental health. Each dimension is scored on a scale from 0 to 100, where 0 represents the worst health status and 100 the best. The SF-36 allows for the calculation of two overall scores: one for physical health and another for mental health.

SECONDARY OUTCOMES:
Visual Analogic Scales (VAS) | At the inclusion of the patient and up to 8 weeks.
  This scale consists of a 10 cm horizontal line, marked at both ends with descriptors such as "not at all" (0) to "completely" (10). Participants are asked to rate their feelings from 0 to 10 regarding four symptoms: "I feel anxious," "I have sleep disturbances," "I have disabling pain," and "I exhibit behavioral disturbances."
State-Trait Anxiety Inventory (STAI) | At the inclusion of the patient and up to 8 weeks
  Anxiety will be evaluated using the State-Trait Anxiety Inventory (STAI). The STAI is a psychometric tool that measures two aspects of anxiety: state anxiety (temporary anxiety related to a specific situation) and trait anxiety (stable, dispositional anxiety). It consists of two subscales, each with 20 items, rated from 1 (not at all) to 4 (very much). The total score for each subscale ranges from 20 to 80, with higher scores indicating higher levels of anxiety.
Questionnaire DysEXecutif (DEX) - Behavioural Assessment of the Dysexecutive Syndrome (BADS) | At the inclusion of the patient and up to 8 weeks
  The severity of behavioral disorders will be assessed using the DEX questionnaire from the Behavioural Assessment of the Dysexecutive Syndrome (BADS). This questionnaire was developed to evaluate executive dysfunction in daily life activities. It is a self-assessment measure consisting of 20 items that assess four dysexecutive criteria: behavioral, cognitive, motivational, and emotional changes, compared to premorbid functioning. Each item is rated on a 5-point Likert scale ranging from "never" to "very often." The sum of each item provides an overall score from 0 to 80. The higher the score, the more severe the executive disorders are. This questionnaire has the advantage of providing both a self-assessment from the patient and an external assessment by the patient's referring neuropsychologist.
Beck Depression Inventory, BDI | At the inclusion of the patient and at up to 8 weeks
  This questionnaire is a self-reported tool consisting of 21 items, each rated from 0 to 3, assessing various symptoms of depression such as mood, cognition, sleep, and appetite. The total score ranges from 0 to 63, with thresholds indicating the severity of depression: 0-13 (minimal depression), 14-19 (mild), 20-28 (moderate), and 29-63 (severe). The scale is commonly used in both clinical practice and research to track the progression of depressive symptoms and measure the effectiveness of treatments.
Pittsburgh Sleep Quality Index (PSQI) | At the inclusion of the patient and up to 8 weeks
  This self-reported questionnaire is designed to assess sleep quality and its impact on health over a 1-month period. It measures 7 components of sleep: subjective quality, sleep onset latency, sleep duration, usual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Each component is rated from 0 to 3, with a total score ranging from 0 to 21. A score higher than 5 indicates poor sleep quality.

OTHER OUTCOMES:
Montreal Cognitive Assessment (MoCA) | At the inclusion of the patient
  The MoCA is a cognitive assessment designed as a quick screening tool for detecting mild cognitive impairment. The MoCA evaluates the following cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructive skills, conceptual thinking, calculations, and spatiotemporal orientation. This scale provides a total score out of 30, which is the sum of the different scores obtained in the sub-scores. With a threshold score of 26, a total score of 26 or higher is considered a normal score. A score below 26 indicates mild cognitive deficits. Investigators choose this scale both for its ease and speed of administration and for its sensitivity to even mild cognitive impairments.
Glasgow Coma Scale (GCS) | At the inclusion of patient
  The GCS is an assessment scale for evaluating the level of consciousness. This scale is a structured evaluation based on 3 components, measured independently: eye opening (E), verbal response (V), and motor response (M). Each sub-scale has a number of grades, starting with the most severe score. Specifically, the "eye opening (E)" sub-scale ranges from 1 (no eye opening) to 4 points (spontaneous eye opening). The "verbal response (V)" sub-scale ranges from 1 (no verbal response) to 5 points (oriented response). Finally, the "motor response (M)" sub-scale ranges from 1 (no motor response) to 6 points (obeys commands). These 3 sub-scales give a total score between 3 (minimum possible score) and 15 (maximum possible score). Regarding interpretation, a score of 15 indicates a normal state. A score between 14 and 10 indicates drowsiness or light coma, while a score between 9 and 4 indicates an increasingly deep coma or unconsciousness. Finally, a score of 3 corresponds to a very deep coma.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Liège, Tinlot, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagendra BD, Ramesh T, Meena M, Study of epidemiology of traumatic brain injury and prevalence of psychiatric disorders in traumatic brain injury at 3 months follow-up, 2019, Nepal Journal of Neurosciences 16 : 8-15.